CLINICAL TRIAL: NCT02153671
Title: Immunogenicity of OrniFlu® Inactivated Influenza Vaccine in Subjects Previously Immunized With Live Attenuated H5N2 Influenza Vaccine and in Non-vaccinated Subjects
Brief Title: Immunogenicity of H5N1 Vaccine Following H5N2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Institute of Experimental Medicine, Russia (Other); Research Institute of Influenza, Russia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LAIV-H5N2-02
Record Dates: First submitted 2014-05-23; First posted 2014-06-03 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Influenza Vaccine
Keywords: LAIV H5N2; Influenza vaccine; Russia
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primed with H5N2 (Experimental): Subjects who received A(H5N1) inactivated influenza vaccine as well as primed with H5N2 live attenuated influenza vaccine approximately 1.5 years before
  Interventions: Biological: A(H5N1) inactivated influenza vaccine (IIV); Biological: A(H5N2) live attenuated influenza vaccine (LAIV)
- Did not receive A(H5N2) (Active Comparator): Subjects who received A(H5N1) inactivated influenza vaccine and did not receive A(H5N2) live attenuated influenza vaccine in a previous study.
  Interventions: Biological: A(H5N1) inactivated influenza vaccine (IIV)

INTERVENTIONS:
Biological: A(H5N1) inactivated influenza vaccine (IIV) — Prepared from the NIBRG-23 vaccine virus strain. One vaccine dose (0.5 ml) contained 15 mg of influenza A(H5N1) virus hemagglutinin (HA), adjuvanted with aluminum hydroxide. Two doses were administered intramuscularly 28 days apart.
  Other Names: Orniflu
Biological: A(H5N2) live attenuated influenza vaccine (LAIV) — Two doses of A(H5N2) live attenuated influenza vaccine (LAIV) administered 28 days apart, approximately 1.5 years prior to receiving A(H5N1) IIV
  Arms: Primed with H5N2

SUMMARY:
This study is designed to assess whether a live attenuated Influenza vaccine (LAIV) can induce a long-lasting immune memory by comparing the immunologic response to two doses of the OrniFlu® inactivated vaccine given to subjects previously primed with LAIV and subjects who did not received LAIV.

DETAILED DESCRIPTION:
This study evaluated immunogenicity of an adjuvanted A(H5N1) inactivated influenza vaccine (IIV) in healthy adult subjects who received A(H5N2) live attenuated influenza vaccine (LAIV) 1.5 years earlier (September/October 2012) and compared this with a group of naive subjects that did not participate in the previous study. Inclusion/exclusion criteria for the additional group of naive volunteers mirrored those utilized in the initial study.

ELIGIBILITY:
Inclusion Criteria:

* Legal male or female adult 18 through 51 years of age at the enrollment visit
* Literate and willing to provide written informed consent
* A signed informed consent
* Free of obvious health problems, as established by the medical history and screening evaluations, including physical examination
* Capable and willing to complete a memory aid and willing to return for all follow-up visits
* For females, willing to take reliable birth control measures through Day 56

Exclusion Criteria:

* Participation in another clinical trial involving any investigational agent within the previous three months or planned enrollment in such a trial during the period of this study
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt
* Participation in any other clinical trials involving any H5-matched influenza vaccines except that in Protocol LAIV-H5N2-01
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever
* Other acute illness at the time of study enrollment
* Receipt of immunoglobulin or other blood products within three months prior to study enrollment or planned receipt during study period
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants and/or immune-modulating therapy within six months prior to study enrollment
* History of bronchial asthma
* Hypersensitivity after previous administration of any (not only influenza) vaccines.
* Other adverse event (AE) following immunization at least possibly related to previous receipt of any (not only influenza) vaccine
* Suspected or known hypersensitivity to any of the study vaccine components, including protein of chicken eggs
* Seasonal (autumnal) hypersensitivity to the natural environment
* Acute or chronic clinically significant abnormality, as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives. Subjects with physical examination findings or clinical laboratory screening results which would be graded 2 or higher on the AE severity grading scale will be excluded from entry into the study
* History of leukemia or any other blood diseases or solid organ cancer
* History of thrombocytopenic purpura or known bleeding disorder
* History of seizures
* Known or suspected immunosuppressive or immunodeficient condition of any kind, including HIV infection
* Known chronic hepatitis B virus (HBV) or hepatitis C (HCV) infection
* Known tuberculosis infection or evidence of previous tuberculosis exposure
* History of chronic alcohol abuse and/or illegal drug use
* Pregnancy or lactation.

  * Systemic connective tissue disorders
* Adrenal gland diseases
* Hereditary, degenerative and progredient diseases of the nervous system
* Any condition that, in the opinion of the investigator, would increase the health risk to the subject if he/she participates in the study or would interfere with the evaluation of the study objectives
* Allergic, including anaphylactic, reactions to any (not only influenza) vaccines

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg I Kiselev, Ph.D., Principal Investigator — Research Institute of Influenza
Locations (1):
- Research Institute of Influenza, Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- H5N2 Primed: Subjects who received A(H5N1) inactivated influenza vaccine as well as A(H5N2) live attenuated influenza vaccine approximately 1.5 years before
  A(H5N1) inactivated influenza vaccine (IIV): Prepared from the NIBRG-23 vaccine virus strain. One vaccine dose (0.5 ml) contained 15 mg of influenza A(H5N1) virus hemagglutinin (HA), adjuvanted with aluminum hydroxide. Two doses were administered intramuscularly 28 days apart.
  A(H5N2) live attenuated influenza vaccine (LAIV): Two doses administered 28 days apart, approximately 1.5 years prior to receiving A(H5N1) IIV
- Control: Subjects who received A(H5N1) inactivated influenza vaccine and did not receive A(H5N2) live attenuated influenza vaccine in a previous study.
  A(H5N1) inactivated influenza vaccine (IIV): Prepared from the NIBRG-23 vaccine virus strain. One vaccine dose (0.5 ml) contained 15 mg of influenza A(H5N1) virus hemagglutinin (HA), adjuvanted with aluminum hydroxide. Two doses were administered intramuscularly 28 days apart.
Period: Overall Study
Arm/Group | H5N2 Primed | Control
Started | 19 | 24
Completed | 19 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | H5N2 Primed | Total
Number analyzed (Participants) | 24 | 19 | 43
Age, Continuous [Mean (Full Range); unit: years] | 30.3 [20 to 48] | 30.8 [20 to 51] | 30.5 [20 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 19 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer of Serum Hemagglutination Inhibition Antibody Response to A/17/Duck/Potsdam/86/92 (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: The following H5 antigens were tested to evaluate the breadth of the response: i) A/17/turkey/Turkey/05/133 (H5N2) (17/t/Tur (H5N2)); ii) A/turkey/Turkey/5/05(H5N1) PR8-based candidate vaccine virus (NIBRG-23 (H5N1)); iii) A/Indonesia/5/2005 (H5N1) PR8-based candidate vaccine virus (Indo (H5N1)); and iv) A/17/duck/Potsdam/86/92 (H5N2) (d/Pot (H5N2)). HAI tests were performed on serum samples with the conventional World Health Organization (WHO)-recommended assays. Sera were pretreated with receptor destroying enzyme (RDE, Denka Seiken, Japan) and tested against 4 HA units of several H5 antigens using horse red blood cells. A four-fold or greater antibody rise in titer was considered to be a seroconversion.
Time Frame: 56 days
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
titer
  Day 0 | 2.7 [2.3 to 3.1] | 2.5 [2.5 to 2.5]
  Day 7 | 7.2 [3.8 to 13.7] | 3.1 [2.4 to 4.2]
  Day 28 | 32.1 [12.8 to 80.5] | 5.9 [3.1 to 11.5]
  Day 56 | 37.2 [15.5 to 89.3] | 9.2 [4.4 to 19.0]

2. Primary Outcome: Geometric Mean Titer of Serum Hemagglutination Inhibition Antibody Response to A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: The following H5 antigens were tested to evaluate the breadth of the response: i) A/17/turkey/Turkey/05/133 (H5N2) (17/t/Tur (H5N2)); ii) A/turkey/Turkey/5/05(H5N1) PR8-based candidate vaccine virus (NIBRG-23 (H5N1)); iii) A/Indonesia/5/2005 (H5N1) PR8-based candidate vaccine virus (Indo (H5N1)); and iv) A/17/duck/Potsdam/86/92 (H5N2) (d/Pot (H5N2)). HAI tests were performed on serum samples with the conventional WHO-recommended assays. Sera were pretreated with receptor destroying enzyme (RDE, Denka Seiken, Japan) and tested against 4 HA units of several H5 antigens using horse red blood cells. A four-fold or greater antibody rise in titer was considered to be a seroconversion.
Time Frame: 56 days
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
titer
  Day 0 | 2.5 [2.5 to 2.5] | 2.5 [2.5 to 2.5]
  Day 7 | 5.2 [2.4 to 11.1] | 3.1 [2.3 to 4.2]
  Day 28 | 43.0 [14.7 to 125.9] | 5.8 [3.1 to 10.8]
  Day 56 | 62.0 [23.3 to 164.9] | 7.1 [3.7 to 13.4]

3. Primary Outcome: Geometric Mean Titer of Serum Hemagglutination Inhibition Antibody Response to A/Indonesia/5/2005 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 2
Time Frame: 56 days
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
titer
  Day 0 | 2.6 [2.4 to 2.8] | 2.6 [2.4 to 3.0]
  Day 7 | 6.5 [3.7 to 11.3] | 3.4 [2.4 to 4.9]
  Day 28 | 35.9 [12.6 to 102.1] | 8.7 [4.4 to 17.2]
  Day 56 | 49.8 [21.2 to 117.2] | 11.9 [5.9 to 23.9]

4. Primary Outcome: Geometric Mean Titer of Serum Hemagglutination Inhibition Antibody Response to A/Turkey/Turkey/5/05(H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 2
Time Frame: 56 days
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
titer
  Day 0 | 2.5 [2.5 to 2.5] | 2.5 [2.5 to 2.5]
  Day 7 | 7.5 [3.0 to 18.5] | 3.1 [2.3 to 4.3]
  Day 28 | 32.1 [10.3 to 100.6] | 5.9 [3.1 to 11.2]
  Day 56 | 44.6 [17.5 to 113.5] | 9.2 [4.7 to 17.8]

5. Primary Outcome: Geometric Mean Titer of Microneutralization Antibody Response to A/17/Turkey/Turkey/05/133 (H5N2) (17/t/Tur (H5N2)) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: Serum specimens were tested for neutralizing antibodies against A/17/turkey/Turkey/05/133 (H5N2) (17/t/Tur (H5N2)) LAIV strain and A/Indonesia/5/2005 (H5N1) PR8-based candidate vaccine virus (Indo (H5N1) by MN using Madin-Darby Canine Kidney cells. Titers of neutralizing antibodies were expressed as reciprocal of the greatest dilution giving a neutralization of 50% on the cytopathic effects of the virus in the tissue culture (TCID50).
Time Frame: 56 days
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
titer
  Day 0 | 14.4 [9.7 to 21.3] | 6.1 [5.3 to 7.0]
  Day 7 | 138.3 [55.7 to 343.1] | 25.2 [12.7 to 49.9]
  Day 28 | 413.1 [205.7 to 829.7] | 58.2 [26.9 to 126.0]
  Day 56 | 370.3 [223.4 to 613.7] | 155.4 [91.0 to 265.5]

6. Primary Outcome: Geometric Mean Titer of Microneutralization Antibody Response to A/Indonesia/5/2005 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 5
Time Frame: 56 days
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
titer
  Day 0 | 8.0 [6.3 to 10.3] | 5.5 [4.9 to 6.0]
  Day 7 | 66.7 [26.8 to 165.7] | 15.9 [9.5 to 26.6]
  Day 28 | 165.9 [83.2 to 331.1] | 31.7 [17.6 to 57.3]
  Day 56 | 239.0 [142.9 to 399.7] | 73.4 [47.1 to 114.2]

7. Primary Outcome: Number and Percentage of Subjects With Seroconversion for Serum Hemagglutination Inhibition (HAI) Antibody Against 17/t/Tur (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: A four-fold or greater antibody rise in titer was considered to be a seroconversion. The following H5 antigens were tested to evaluate the breadth of the response: i) A/17/turkey/Turkey/05/133 (H5N2) (17/t/Tur (H5N2)); ii) A/turkey/Turkey/5/05(H5N1) PR8-based candidate vaccine virus (NIBRG-23 (H5N1)); iii) A/Indonesia/5/2005 (H5N1) PR8-based candidate vaccine virus (Indo (H5N1)); and iv) A/17/duck/Potsdam/86/92 (H5N2) (d/Pot (H5N2)). HAI tests were performed on serum samples with the conventional WHO-recommended assays. Sera were pretreated with receptor destroying enzyme (RDE, Denka Seiken, Japan) and tested against 4 HA units of several H5 antigens using horse red blood cells.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroconversion | 5 | 2
  Day 7: No seroconversion | 14 | 22
  Day 28: Seroconversion | 13 | 6
  Day 28: No seroconversion | 6 | 18
  Day 56: Seroconversion | 15 | 10
  Day 56: No seroconversion | 4 | 14

8. Primary Outcome: Number and Percentage of Subjects With Seroconversion for Serum Hemagglutination Inhibition (HAI) Antibody Against A/Turkey/Turkey/5/05 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 7
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroconversion | 5 | 2
  Day 7: No seroconversion | 14 | 22
  Day 28: Seroconversion | 11 | 7
  Day 28: No seroconversion | 8 | 17
  Day 56: Seroconversion | 14 | 12
  Day 56: No seroconversion | 5 | 12

9. Primary Outcome: Number and Percentage of Subjects With Seroconversion for Serum Hemagglutination Inhibition (HAI) Antibody Against A/Indonesia/5/2005 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 7
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroconversion | 8 | 2
  Day 7: No seroconversion | 11 | 22
  Day 28: Seroconversion | 12 | 10
  Day 28: No seroconversion | 7 | 14
  Day 56: Seroconversion | 15 | 13
  Day 56: No seroconversion | 4 | 11

10. Primary Outcome: Number and Percentage of Subjects With Seroconversion for Serum Hemagglutination Inhibition (HAI) Antibody Against A/17/Duck/Potsdam/86/92 (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 7
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroconversion | 7 | 3
  Day 7: No seroconversion | 12 | 21
  Day 28: Seroconversion | 14 | 7
  Day 28: No seroconversion | 5 | 17
  Day 56: Seroconversion | 14 | 10
  Day 56: No seroconversion | 5 | 14

11. Primary Outcome: Number and Percentage of Subjects With Seroconversion for Microneutralization (MN) Antibody Against A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: Serum specimens were tested for neutralizing antibodies against A/17/turkey/Turkey/05/133 (H5N2) (17/t/Tur (H5N2)) LAIV strain and A/Indonesia/5/2005 (H5N1) PR8-based candidate vaccine virus (Indo (H5N1) by MN using Madin-Darby Canine Kidney cells. Titers of neutralizing antibodies were expressed as reciprocal of the greatest dilution giving a neutralization of 50% on the cytopathic effects of the virus in the tissue culture (TCID50). A four-fold or greater antibody rise in titer was considered to be a seroconversion.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroconversion | 12 | 11
  Day 7: No seroconversion | 7 | 13
  Day 28: Seroconversion | 18 | 18
  Day 28: No seroconversion | 1 | 6
  Day 56: Seroconversion | 18 | 23
  Day 56: No seroconversion | 1 | 1

12. Primary Outcome: Number and Percentage of Subjects With Seroconversion for Microneutralization (MN) Antibody Against A/Indonesia/5/2005 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 11
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroconversion | 11 | 11
  Day 7: No seroconversion | 8 | 13
  Day 28: Seroconversion | 18 | 16
  Day 28: No seroconversion | 1 | 8
  Day 56: Seroconversion | 19 | 23
  Day 56: No seroconversion | 0 | 1

13. Primary Outcome: Number and Percentage of Subjects With Seroprotective Titers for Serum Hemagglutination Inhibition (HAI) Antibody Against 17/t/Tur (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: Seroprotection was defined as ≥1:40 antibody titer. The following H5 antigens were tested to evaluate the breadth of the response: i) A/17/turkey/Turkey/05/133 (H5N2) (17/t/Tur (H5N2)); ii) A/turkey/Turkey/5/05(H5N1) PR8-based candidate vaccine virus (NIBRG-23 (H5N1)); iii) A/Indonesia/5/2005 (H5N1) PR8-based candidate vaccine virus (Indo (H5N1)); and iv) A/17/duck/Potsdam/86/92 (H5N2) (d/Pot (H5N2)). HAI tests were performed on serum samples with the conventional WHO-recommended assays. Sera were pretreated with receptor destroying enzyme (RDE, Denka Seiken, Japan) and tested against 4 HA units of several H5 antigens using horse red blood cells.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroprotection | 4 | 1
  Day 7: No seroprotection | 15 | 23
  Day 28: Seroprotection | 11 | 3
  Day 28: No seroprotection | 8 | 21
  Day 56: Seroprotection | 14 | 7
  Day 56: No seroprotection | 5 | 17

14. Primary Outcome: Number and Percentage of Subjects With Seroprotective Titer of Serum Hemagglutination Inhibition (HAI) Antibody Against A/Turkey/Turkey/5/05 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 13
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroprotection | 5 | 1
  Day 7: No seroprotection | 14 | 23
  Day 28: Seroprotection | 11 | 3
  Day 28: No seroprotection | 8 | 21
  Day 56: Seroprotection | 14 | 7
  Day 56: No seroprotection | 5 | 17

15. Primary Outcome: Number and Percentage of Subjects With Seroprotective Titer of Serum Hemagglutination Inhibition (HAI) Antibody Against A/Indonesia/5/2005 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 13
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroprotection | 2 | 2
  Day 7: No seroprotection | 17 | 22
  Day 28: Seroprotection | 12 | 4
  Day 28: No seroprotection | 7 | 20
  Day 56: Seroprotection | 14 | 9
  Day 56: No seroprotection | 5 | 15

16. Primary Outcome: Number and Percentage of Subjects With Seroprotective Titer of Serum Hemagglutination Inhibition (HAI) Antibody Against A/17/Duck/Potsdam/86/92 (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 13
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroprotection | 5 | 1
  Day 7: No seroprotection | 14 | 23
  Day 28: Seroprotection | 11 | 4
  Day 28: No seroprotection | 8 | 20
  Day 56: Seroprotection | 14 | 8
  Day 56: No seroprotection | 5 | 16

17. Primary Outcome: Number and Percentage of Subjects With Seroprotective Titer of Microneutralization (MN) Antibody Against A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: Serum specimens were tested for neutralizing antibodies against A/17/turkey/Turkey/05/133 (H5N2) (17/t/Tur (H5N2)) LAIV strain and A/Indonesia/5/2005 (H5N1) PR8-based candidate vaccine virus (Indo (H5N1) by MN using Madin-Darby Canine Kidney cells. Titers of neutralizing antibodies were expressed as reciprocal of the greatest dilution giving a neutralization of 50% on the cytopathic effects of the virus in the tissue culture (TCID50). Seroprotection was defined as ≥1:40 antibody titer.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroprotection | 15 | 7
  Day 7: No seroprotection | 4 | 17
  Day 28: Seroprotection | 19 | 14
  Day 28: No seroprotection | 0 | 10
  Day 56: Seroprotection | 19 | 22
  Day 56: No seroprotection | 0 | 2

18. Primary Outcome: Number and Percentage of Subjects With Seroprotective Titer of Microneutralization (MN) Antibody Against A/Indonesia/5/2005 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 17
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroprotection | 12 | 6
  Day 7: No seroprotection | 7 | 18
  Day 28: Seroprotection | 17 | 11
  Day 28: No seroprotection | 2 | 13
  Day 56: Seroprotection | 19 | 21
  Day 56: No seroprotection | 0 | 3

19. Primary Outcome: Geometric Mean Titer of Serum Immunoglobulin A (IgA) Response to A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: Detection of anti-hemagglutinin (HA) immunoglobulin A (IgA) and immunoglobulin G (IgG) antibodies was carried out by indirect enzyme-linked immunosorbent assay (ELISA). 16 HA units of sucrose-purified virus antigen was used to coat ELISA plates in a volume of 100 ml. Two-fold dilutions of sera were prepared starting from 1:10 (for IgA antibody) and 1:100 (for IgG antibody) and added to the coated wells, followed by incubation with the horseradish peroxidase-conjugated goat anti-human IgA or IgG.
Time Frame: 56 days
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
titer
  Day 0 | 4.5 (1.4) | 4.0 (1.7)
  Day 7 | 6.2 (1.9) | 5.0 (1.4)
  Day 28 | 6.8 (1.5) | 5.3 (1.5)
  Day 56 | 6.7 (1.4) | 5.2 (1.7)

20. Primary Outcome: Geometric Mean Titer of Serum Immunoglobulin A (IgA) Response to A/Turkey/Turkey/5/05 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 19
Time Frame: 56 days
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
titer
  Day 0 | 2.5 (0.8) | 2.5 (1.2)
  Day 7 | 5.3 (2.4) | 4.1 (1.5)
  Day 28 | 5.6 (2.3) | 3.9 (2.1)
  Day 56 | 5.6 (1.9) | 4.2 (2.1)

21. Primary Outcome: Geometric Mean Titer of Serum Immunoglobulin G (IgG) Response to A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 19
Time Frame: 56 days
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
titer
  Day 0 | 9.7 (0.9) | 9.0 (1.1)
  Day 7 | 10.4 (1.1) | 9.7 (1.2)
  Day 28 | 11.2 (1.1) | 10.2 (1.3)
  Day 56 | 11.3 (0.9) | 10.6 (1.0)

22. Primary Outcome: Geometric Mean Titer of Serum Immunoglobulin G (IgG) Response to A/Turkey/Turkey/5/05 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 19
Time Frame: 56 days
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
titer
  Day 0 | 8.3 (1.1) | 9.5 (1.1)
  Day 7 | 10.4 (1.1) | 9.7 (1.2)
  Day 28 | 11.2 (1.1) | 10.2 (1.3)
  Day 56 | 10.3 (0.9) | 9.2 (1.3)

23. Primary Outcome: Number and Percentage of Subjects With Seroconversion for Immunoglobulin A (IgA) Against A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: A four-fold or greater antibody rise in titer was considered to be a seroconversion. Detection of anti-hemagglutinin (HA) immunoglobulin A (IgA) and immunoglobulin G (IgG) antibodies was carried out by indirect enzyme-linked immunosorbent assay (ELISA). 16 HA units of sucrose-purified virus antigen was used to coat ELISA plates in a volume of 100 ml. Two-fold dilutions of sera were prepared starting from 1:10 (for IgA antibody) and 1:100 (for IgG antibody) and added to the coated wells, followed by incubation with the horseradish peroxidase-conjugated goat anti-human IgA or IgG.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroconversion | 9 | 8
  Day 7: No seroconversion | 10 | 16
  Day 28: Seroconversion | 13 | 9
  Day 28: No seroconversion | 6 | 15
  Day 56: Seroconversion | 13 | 9
  Day 56: No seroconversion | 6 | 15

24. Primary Outcome: Number and Percentage of Subjects With Seroconversion for Immunoglobulin A (IgA) Against A/Turkey/Turkey/5/05 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 23
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroconversion | 15 | 12
  Day 7: No seroconversion | 4 | 12
  Day 28: Seroconversion | 15 | 11
  Day 28: No seroconversion | 4 | 13
  Day 56: Seroconversion | 15 | 13
  Day 56: No seroconversion | 4 | 11

25. Primary Outcome: Number and Percentage of Subjects With Seroconversion for Immunoglobulin G (IgG) Against A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 23
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroconversion | 3 | 4
  Day 7: No seroconversion | 16 | 20
  Day 28: Seroconversion | 9 | 7
  Day 28: No seroconversion | 10 | 17
  Day 56: Seroconversion | 10 | 10
  Day 56: No seroconversion | 9 | 14

26. Primary Outcome: Number and Percentage of Subjects With Seroconversion for Immunoglobulin G (IgG) Against A/Turkey/Turkey/5/05 (H5N1) PR8-based Candidate Vaccine Virus Following Administration of A(H5N1) Inactivated Influenza Vaccine (IIV)
Description: as for outcome 23
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: Seroconversion | 5 | 6
  Day 7: No seroconversion | 14 | 18
  Day 28: Seroconversion | 11 | 11
  Day 28: No seroconversion | 8 | 13
  Day 56: Seroconversion | 11 | 15
  Day 56: No seroconversion | 8 | 9

27. Secondary Outcome: Number and Percentage of Subjects With ≥15% Increase of Avidity Index in Serum Immunoglobulin A (IgA) Against A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain After Receiving One Dose of A(H5N1) Inactivated Influenza Vaccine
Description: The avidity index (AI) was defined as the ratio of the mean optical density at 450 nm (OD450) with urea to that without urea, multiplied by 100. A 15% increase in the AI value was considered significant.
Time Frame: 28 days
Population: Subjects with seroconversion were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Day 7: number analyzed (Participants) | 14 | 9
  Day 7: Yes | 6 | 2
  Day 7: No | 8 | 7
  Day 28: number analyzed (Participants) | 14 | 9
  Day 28: Yes | 5 | 1
  Day 28: No | 9 | 8

28. Secondary Outcome: Number and Percentage of Subjects With ≥15% Increase of Avidity Index in Serum Immunoglobulin G (IgG) Against A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain After Receiving One Dose of A(H5N1) Inactivated Influenza Vaccine
Description: as for outcome 27
Time Frame: 28 days
Population: Subjects with seroconversion were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 11 | 11
Participants
  Day 7: Yes | 5 | 1
  Day 7: No | 6 | 10
  Day 28: Yes | 6 | 1
  Day 28: No | 5 | 10

29. Secondary Outcome: Number and Percentage of Subjects With ≥15% Increase of Avidity Index in Serum Immunoglobulin A (IgA) Against A/Turkey/Turkey/5/05 (H5N1) PR8-based Candidate Vaccine Virus After Receiving One Dose of A(H5N1) Inactivated Influenza Vaccine
Description: as for outcome 27
Time Frame: 28 days
Population: Subjects with seroconversion were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 17 | 16
Participants
  Day 7: Yes | 9 | 3
  Day 7: No | 8 | 13
  Day 28: Yes | 7 | 0
  Day 28: No | 10 | 16

30. Secondary Outcome: Number and Percentage of Subjects With ≥15% Increase of Avidity Index in Serum Immunoglobulin G (IgG) Against A/Turkey/Turkey/5/05 (H5N1) PR8-based Candidate Vaccine Virus After Receiving One Dose of A(H5N1) Inactivated Influenza Vaccine
Description: as for outcome 27
Time Frame: 28 days
Population: Subjects with seroconversion were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 11 | 17
Participants
  Day 7: Yes | 2 | 0
  Day 7: No | 9 | 17
  Day 28: Yes | 6 | 3
  Day 28: No | 5 | 14

31. Secondary Outcome: Mean Avidity Index for Serum Immunoglobulin A (IgA) Against A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain After Receiving One Dose of A(H5N1) Inactivated Influenza Vaccine
Description: as for outcome 27
Time Frame: 28 days
Population: Subjects with seroconversion were included in the analysis.
Measure: Mean (Standard Deviation); unit: avidity index
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 14 | 9
avidity index
  Day 0 | 75.6 (14.6) | 75.2 (8.6)
  Day 7 | 87.7 (9.3) | 81.5 (10.3)
  Day 28 | 87.2 (8.6) | 85.1 (7.8)

32. Secondary Outcome: Mean Avidity Index for Serum Immunoglobulin G (IgG) Against A/17/Turkey/Turkey/05/133 (H5N2) LAIV Strain After Receiving One Dose of A(H5N1) Inactivated Influenza Vaccine
Description: as for outcome 27
Time Frame: 28 days
Population: Subjects with seroconversion were included in the analysis.
Measure: Mean (Standard Deviation); unit: avidity index
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 11 | 11
avidity index
  Day 0 | 81.6 (11.8) | 83.4 (9.7)
  Day 7 | 90.7 (5.7) | 86.0 (12.0)
  Day 28 | 92.3 (6.4) | 84.2 (10.5)

33. Secondary Outcome: Mean Avidity Index for Serum Immunoglobulin A (IgA) Against A/Turkey/Turkey/5/05 (H5N1) PR8-based Candidate Vaccine Virus After Receiving One Dose of A(H5N1) Inactivated Influenza Vaccine
Description: as for outcome 27
Time Frame: 28 days
Population: Subjects with seroconversion were included in the analysis.
Measure: Mean (Standard Deviation); unit: avidity index
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 17 | 16
avidity index
  Day 0 | 72.7 (7.5) | 77.4 (6.4)
  Day 7 | 86.4 (12.6) | 83.3 (8.1)
  Day 28 | 84.9 (8.8) | 77.9 (8.3)

34. Secondary Outcome: Mean Avidity Index for Serum Immunoglobulin G (IgG) Against A/Turkey/Turkey/5/05 (H5N1) PR8-based Candidate Vaccine Virus After Receiving One Dose of A(H5N1) Inactivated Influenza Vaccine
Description: as for outcome 27
Time Frame: 28 days
Population: Subjects with seroconversion were included in the analysis.
Measure: Mean (Standard Deviation); unit: avidity index
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 11 | 17
avidity index
  Day 0 | 76.2 (4.9) | 78.3 (8.2)
  Day 7 | 86.2 (10.6) | 78.0 (9.1)
  Day 28 | 90.6 (14.2) | 77.9 (15.8)

35. Other Pre Specified Outcome: Number of Subjects Experiencing Adverse Events After Receiving A(H5N1) Inactivated Influenza Vaccine
Description: Subjects were asked to closely watch for and report any adverse events occurring the first 6 days after immunization, and followed for any reactions and adverse events occurring within 7 and 28 days after each vaccination.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Post-dose 1: Mild | 13 | 14
  Post-dose 1: Moderate | 0 | 1
  Post-dose 1: None | 6 | 9
  Post-dose 2: Mild | 9 | 3
  Post-dose 2: Moderate | 1 | 1
  Post-dose 2: None | 9 | 20

36. Other Pre Specified Outcome: Number of Subjects Experiencing Any Adverse Event Related to the A(H5N1) Inactivated Influenza Vaccine
Description: as for outcome 35
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | H5N2 Primed | Control
Number analyzed (Participants) | 19 | 24
Participants
  Post-dose 1: Experienced treatment-related adverse event | 11 | 9
  Post-dose 1: Did not experience treatment-related adverse event | 8 | 15
  Post-dose 2: Experienced treatment-related adverse event | 9 | 4
  Post-dose 2: Did not experience treatment-related adverse event | 10 | 20

ADVERSE EVENTS:
Time Frame: 56 days
Description: Subjects were asked to closely watch for and report any adverse events occurring the first 6 days after immunization, and followed for any reactions and adverse events occurring within 7 and 28 days after each vaccination
Arm/Group | H5N2 Primed | Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/24
Other Adverse Events (participants affected / at risk) | 17/19 | 15/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | H5N2 Primed (N=19) | Control (N=24)
Headache (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Bilirubin increased (Investigations) | 0 | 4
Blood creatinine increased (Investigations) | 3 | 1
Eosinophil count increased (Investigations) | 8 | 4
Lymphocyte count increased (Investigations) | 5 | 1
Lymphocyte count decreased (Investigations) | 8 | 6
Monocyte count increased (Investigations) | 4 | 5
Neutrophil count increased (Investigations) | 7 | 8
Neutrophil count decreased (Investigations) | 7 | 8
White blood cells count increased (Investigations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No